CLINICAL TRIAL: NCT04066595
Title: Cabozantinib in Patients With Locally Advanced or Metastatic Urothelial Cell Carcinoma Who Have Progressed After Cisplatin-based Chemotherapy and Anti-PD-1/PD-L1 Therapy or After Anti-PD-1/PD-L1 Therapy Only.
Brief Title: Cabozantinib in Patients With Locally Advanced or Metastatic Urothelial Cell Carcinoma.
Acronym: CabUC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Interdisciplinary Center Clinical Trials (IZKS), University Medical Center Mainz (Unknown)
Responsible Party: Principal Investigator, Georg Bartsch, Assistant Medical Director of Department of Urology and Pediatric Urology, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CabUC
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: 2 cohorts. Cohort 1 will consist of patients who have been pre-treated with checkpoint inhibitors only (2nd line setting for cabozantinib). Cohort 2 will consist of patients who have been pre-treated with cisplatin-based chemotherapy and checkpoint inhibitors (3rd line setting for cabozantinib).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (cohorts 1 and 2) (Experimental): Cohort 1 will consist of patients who have been pre-treated with checkpoint inhibitors only (2nd line setting for cabozantinib). Cohort 2 will consist of patients who have been pre-treated with cisplatin-based chemotherapy and checkpoint inhibitors (3rd line setting for cabozantinib). Both cohorts receive the same treatment.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — 60 mg cabozantinib oral daily. When dose reduction is necessary, it is recommended to reduce to 40 mg daily, and then to 20 mg daily.
  Other Names: Cabometyx

SUMMARY:
In this Phase II study we investigate the benefit of cabozantinib treatment for patients with locally advanced or metastasized urothelial cell carcinoma who have been pre-treated with checkpoint inhibitors only (cohort 1) or who have been pre-treated with cisplatin-based chemotherapy and checkpoint inhibitors (cohort 2). We are lacking adequate response and outcome data in patients after immunotherapy and consider that this study will improve future treatment modalities for this important patient cohort.

ELIGIBILITY:
Inclusion criteria:

1. Ability of subject to understand nature, importance and individual consequences of clinical trial.
2. Signed and dated informed consent of the subject must be available before start of any specific trial procedures.
3. Male or female patients ≥ 18 years
4. Life expectancy ≥ 10 weeks, by judgment of the Investigator.
5. Patients must be able to swallow intact tablets.
6. Patients with histology/cytology confirmed urothelial carcinoma (UC) including mixed pathology with predominantly UC, with locally advanced (T4b) or metastatic (lymph node or visceral) UC arising from bladder or upper urinary tracts. Patients with measurable disease (at least one tumor lesion measurable on radiographic imaging as defined by RECIST 1.1).
7. ECOG (Eastern Cooperative Oncology Group) Performance Status 0-1.
8. Cohort 1: patients who have been pre-treated with checkpoint inhibitors only for one of the following reasons: glomerular filtration rate more ≥30 ml/min and ≤ 60 ml/min (Cockcroft-Gault formula), grade 2 or higher hearing loss or peripheral neuropathy. Cohort 2: patients who have been pre-treated with cisplatin-based chemotherapy and checkpoint inhibitors.
9. Recurrence within 12 months (by RECIST criteria version 1.1) from last cycle of chemotherapy or PD-1/PD-L1 therapy.
10. Recovery to baseline or ≤ Grade 1 CTCAE v.5.0 from toxicities related to any prior treatments, unless the side effects are clinically non-significant and/or stable on supportive therapy.

Exclusion criteria:

1. Radiation, chemotherapy, or other anti-cancer therapy < 4 weeks prior to enrollment in the study.
2. Patients previously treated with small molecule tyrosine kinase inhibitors.
3. Systemic treatment with radionuclides < 4 weeks prior to enrollment in the study, and subjects with clinically relevant ongoing complications from prior radiation therapy.
4. Abdominal surgery <10 weeks prior to enrollment in the study. Complete wound healing must be observed at least 10 days prior to enrollment, and patients should not have relevant ongoing complications at study enrollment.
5. Inadequate organ and bone marrow function as evidenced by:

   1. Hemoglobin <9.0 g/dL;
   2. HbA1c > 8%;
   3. Absolute neutrophil count <1.5 x 109/L;
   4. Platelet count <100 x 109/L;
   5. Fasting serum triglycerides > 2.5 x ULN and total cholesterol > 300 mg/dL. Lipid-lowering medication is allowed;
   6. AST (aspartate aminotransferase) /SGOT (serum glutamate oxaloacetate transaminase) and/or ALT (alanine aminotransferase)/SGPT (serum glutamate pyruvate transaminase) ≥3.0 x ULN (upper limit of normal);
   7. Total bilirubin >1.5 x ULN (upper limit of normal), for subjects with Gilbert's disease > 3 mg/dL;
   8. Serum creatinine >2.0 x ULN;
   9. Creatinine clearance ≤ 30 mL/min (Cockroft-Gault formula);
   10. PT (prothrombin time) or INR (international normalized ratio) or PTT (partial thromboplastin time) ≥ 1.3 x ULN.
   11. Urine protein-to-creatinine ratio (UPCR) > 1 mg/mg (> 113.2 mg/mmol)
6. Symptomatic brain metastases or leptomeningeal disease (in case of clinical suspicion of central nervous system involvement confirmed by existing CT or MRI scan of the brain).
7. History of another neoplasm except non-metastatic melanoma skin cancers, carcinoma in situ of the cervix, treated patients with incidental prostate cancer (pT2 (after RPE), Gleason ≤ 6) and PSA (prostate specific antigen) ≤ 0.5 ng/mL, or cancer cured by surgery, small field radiation or chemotherapy <5 years prior to enrollment.
8. History of inflammatory bowel disease, significant bowel obstruction, GI disorder with a high risk of perforation or fistula.
9. Any of the following events within 6 months prior to inclusion: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft surgery, clinically symptomatic and uncontrolled cardiovascular disease, or clinically significant arrhythmias (grade 3-4).
10. Concurrent treatment with strong inhibitors of cytochrome P450 3A4 (including but not limited to cyclosporin, erythromycin, ketoconazole, itraconazole, quinidine, phenobarbital salt with quinidine, ritonavir, valspodar, verapamil, St John's wort, rifampicin) or patients planning to receive these treatments. For patients who were receiving treatment with such agents, a one-week washout period is required prior to enrollment.
11. Currently receiving any other investigational agent or received an investigational agent within 30 days (or within 5 times the half-life of this agent) before the first dose of cabozantinib.
12. Significant allergy to a pharmaceutical therapy that, in the opinion of the Investigator, poses an increased risk to the patient.
13. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
14. Active substance abuse (including active alcohol abuse).
15. Medical or psychological conditions that would jeopardize an adequate and orderly completion of the trial.
16. Women who are pregnant or breastfeeding.
17. Women of childbearing potential (WOCBP, a woman is considered of childbearing potential i.e. fertile, following menarche and until becoming post-menopausal (defined as spontaneous amenorrhea for at least a year) or permanently sterilized (e.g. bilateral oophorectomy, hysterectomy, bilateral salpingectomy)), unless they have a negative serum or urine pregnancy test within 7 days prior to first dose of cabozantinib. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG (human chorionic gonadotropin).
18. Women of childbearing potential, unless they agree to practice a highly effective and medically accepted contraception method during trial and for 4 months after last dose of study drug. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:

    1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

       * oral
       * intravaginal
       * transdermal
    2. progestogen-only hormonal contraception associated with inhibition of ovulation:

       * oral
       * injectable
       * implantable
    3. intrauterine device (IUD)
    4. intrauterine hormone-releasing system (IUS)
    5. bilateral tubal occlusion
    6. vasectomized partner (medical assessment must be present and done)
    7. sexual abstinence when this is in line with the preferred and usual lifestyle of the subject
19. Sexually active male subjects, unless they agree to use contraception (condom, contraception for non-pregnant WOCBP partner) with their partners throughout the study and for 4 months after last dose of study drug and agree to inform the Investigator if the respective partner becomes pregnant during this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate after 6 months of cabozantinib treatment | 6 months
  The response rate is defined as the percentage of subjects with a confirmed reduction in tumor size compared to baseline as well as fulfilling the criteria for complete or partial response according to RECIST 1.1. The response to treatment is measured by computer tomography (CT) every 12 weeks starting from the first day of cabozantinib treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, up to approximately 2 years
  PFS is defined as the time from first intake of trial medication to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm.
1-year survival | 1 year
  Rate of subjects surviving for at least one year after first intake/dose of trial medication
Overall survival | Through study completion, up to approximately 2 years
  The time between first application of trial medication to date of death due to any cause
Clinical benefit rate | Through study completion, up to approximately 2 years
  Complete or partial response or stable disease for ≥ 6 months according to RECIST 1.1
Response duration | Through study completion, up to approximately 2 years
  Duration of response in months from the first response (CR or PR) to progress after first intake of treatment medication
Number of Participants with Adverse Events (AEs) | Through study completion, up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs) | Through study completion, up to approximately 2 years
  The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology of the University Medical Center Mainz, Mainz, Germany